CLINICAL TRIAL: NCT05349630
Title: Impact of Iron Supplementation on Right Ventricular Function and Exercise Performance in Hypoxia (A Sub-Study)
Brief Title: Impact of Iron Supplementation on Right Ventricular Function and Exercise Performance in Hypoxia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 21-4354b
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Right Ventricular Dysfunction; Hypoxia
MeSH Terms: conditions — Ventricular Dysfunction, Right; Hypoxia | interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: All participants will complete resting echocardiography and exercise testing as part of parent study prior to oral iron supplementation. Participants who enroll in this study will complete 30 days of oral iron supplementation and then repeat resting echocardiography and exercise testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy individuals - pre-iron (Placebo Comparator): Five healthy participants will be enrolled. Baseline echocardiography and exercise data prior to oral iron supplementation will be obtained as part of the "parent" study to this study (NCT05272514).
  Interventions: Drug: Ferrous sulfate 325mg
- Healthy individuals - post-iron (Active Comparator): The same five healthy participants will complete echocardiography and exercise testing after taking 30 days of oral iron supplementation.
  Interventions: Drug: Ferrous sulfate 325mg

INTERVENTIONS:
Drug: Ferrous sulfate 325mg — Participants will take one tab of ferrous sulfate 325 mg (equivalent to 65 mg elemental iron) daily for 30 days.

SUMMARY:
The purpose of this study is to determine if taking iron supplement pills improves exercise performance in low-oxygen conditions.

DETAILED DESCRIPTION:
Hypoxia (low oxygen) causes the blood vessels in the lungs to constrict (hypoxic pulmonary vasoconstriction). This increases the pressure (afterload) the right ventricle faces as it pumps blood to the lungs. Increased right ventricular afterload during hypoxia may compromise exercise capacity. Intravenous iron administration prior to hypoxic exposure has been shown to blunt the hypoxia-induced increase in right ventricular afterload. This may be through iron's action in the Hypoxia Inducible Factor (HIF) pathway. Iron is a cofactor for prolyl hydroxylases that degrade HIF subunits and thus may "turn off" HIF-related pathways of pulmonary artery vasoconstriction and remodeling. However, it is not known whether oral iron supplementation similarly reduces right ventricular afterload in hypoxia, or what impact iron has on right ventricular function and exercise capacity in hypoxia.

This is a human physiology study that will characterize the impact of oral iron supplementation on right ventricular function and exercise performance in hypoxia. It is a follow-up "sub-study" to a separate, "parent" study (NCT05272514) by the same investigators which evaluates resting and exertional right ventricular performance in normoxia and hypoxia in 10 healthy individuals. In this follow-up study, 5 individuals who completed the parent study will be eligible to enroll. As part of the parent study, participants will complete baseline echocardiography to assess right ventricular function and cardiopulmonary exercise testing to assess exercise performance in normoxia and hypoxia. After enrolling in this study, participants will take an oral iron supplement (ferrous sulfate 325 mg oral daily) for 30 days. They will then return for one visit. First, participants will complete submaximal exercise while breathing room air. Submaximal exercise will include 5 minutes each at 40% and 60% of baseline hypoxic (fraction of inspired oxygen [FiO2] 12%) maximal oxygen uptake (VO2max) achieved during parent study. After 10 minutes' rest, echocardiographic measurements will be obtained at upright rest with FiO2 21%, 17%, 15%, and 12% to characterize the impact of progressive hypoxia on resting right ventricular function. Participants will then repeat submaximal exercise tests at FiO2 12%, followed by a short period of recovery. Thereafter, participants will complete a symptom-limited cardiopulmonary exercise test at FiO2 12%. Measurements will include heart rate/rhythm, oxygen saturation, blood pressure, gas exchange parameters (oxygen uptake [VO2], carbon dioxide production [VCO2], and minute ventilation), rated perceived exertion and resting echocardiographic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60
* For women, premenopausal status

Exclusion Criteria:

* Active cardiovascular or pulmonary disease (e.g. hypertension, coronary artery disease, cardiomyopathy, arrhythmia, valvular abnormalities, diabetes, peripheral vascular disease, tobacco use, chronic obstructive pulmonary disease, asthma, interstitial lung disease, restrictive lung disease, or pulmonary hypertension)
* Use of cardiac- or pulmonary-related medications
* Prior history of high altitude pulmonary edema or high altitude cerebral edema
* Body mass index < 18.5 or > 30
* Anemia
* Iron deficiency
* Iron supplementation (oral or intravenous) in the preceding 60 days
* Systemic anticoagulation or aspirin use that cannot be temporarily held for the study
* Pregnancy
* Non-cardiopulmonary disorders that adversely influence exercise ability (e.g. arthritis or peripheral vascular disease)
* Dedicated athletic training (defined here as spending >9 hours per week in vigorous physical activity [≥6 mets])
* Regular high-altitude exercise (defined here as engaging in vigorous physical activity [≥1 hour at ≥6 mets] at ≥8,000 ft for >2 days per week over the preceding 4 weeks)
* Residence at ≥8,000 ft for 3 or more consecutive nights in the preceding 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Maximum workload | Up to 1 hour
  Workload in Watts at peak exercise on upright cycle ergometer
Maximal oxygen uptake | Up to 1 hour
  Maximal oxygen uptake at peak exercise (VO2max) in L/min

SECONDARY OUTCOMES:
Oxygen saturation at peak exercise | Up to 1 hour
  Peripheral oxygen saturation (SpO2)
Submaximal Stage 1 workload | Up to 1 hour
  Workload in Watts at 40% x hypoxic VO2max (obtained during baseline hypoxic exercise test)
Submaximal Stage 2 workload | Up to 1 hour
  Workload in Watts at 60% x hypoxic VO2max (obtained during baseline hypoxic exercise test)
Ventilatory threshold | Up to 1 hour
  Oxygen uptake (VO2 in L/min) at which slope of VCO2/VO2 relationship increases
Tricuspid annular plane systolic excursion measured by echocardiography | Up to 1 hour
  In mm
Pulmonary artery systolic pressure measured by echocardiography | Up to 1 hour
  In mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith TG, Balanos GM, Croft QP, Talbot NP, Dorrington KL, Ratcliffe PJ, Robbins PA. The increase in pulmonary arterial pressure caused by hypoxia depends on iron status. J Physiol. 2008 Dec 15;586(24):5999-6005. doi: 10.1113/jphysiol.2008.160960. Epub 2008 Oct 27. PMID 18955380
- [Background] Smith TG, Talbot NP, Privat C, Rivera-Ch M, Nickol AH, Ratcliffe PJ, Dorrington KL, Leon-Velarde F, Robbins PA. Effects of iron supplementation and depletion on hypoxic pulmonary hypertension: two randomized controlled trials. JAMA. 2009 Oct 7;302(13):1444-50. doi: 10.1001/jama.2009.1404. PMID 19809026
- [Background] Cornwell WK, Tran T, Cerbin L, Coe G, Muralidhar A, Hunter K, Altman N, Ambardekar AV, Tompkins C, Zipse M, Schulte M, O'Gean K, Ostertag M, Hoffman J, Pal JD, Lawley JS, Levine BD, Wolfel E, Kohrt WM, Buttrick P. New insights into resting and exertional right ventricular performance in the healthy heart through real-time pressure-volume analysis. J Physiol. 2020 Jul;598(13):2575-2587. doi: 10.1113/JP279759. Epub 2020 May 18. PMID 32347547
- [Background] Cornwell WK 3rd, Baggish AL, Bhatta YKD, Brosnan MJ, Dehnert C, Guseh JS, Hammer D, Levine BD, Parati G, Wolfel EE; American Heart Association Exercise, Cardiac Rehabilitation, and Secondary Prevention Committee of the Council on Clinical Cardiology; and Council on Arteriosclerosis, Thrombosis and Vascular Biology. Clinical Implications for Exercise at Altitude Among Individuals With Cardiovascular Disease: A Scientific Statement From the American Heart Association. J Am Heart Assoc. 2021 Oct 5;10(19):e023225. doi: 10.1161/JAHA.121.023225. Epub 2021 Sep 9. PMID 34496612